CLINICAL TRIAL: NCT02576366
Title: Phenotypic Drug Probes as Predictors of Drug-drug Interactions With Tacrolimus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TacDDI151010
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Drug Interactions; Kidney Transplantation
MeSH Terms: interventions — Voriconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Voriconazole (Experimental): Four hundred mg of voriconazole (2 tablets of 200 mg Vfend; Pfizer, Karlsruhe, Germany) will be administered twice daily on day 2. Two hundred mg of voriconazole (1 tablet of 200 mg Vfend) will be administered twice daily on days 3, 4, 5 and 6.
  Interventions: Drug: Voriconazole
- Rifampin (Experimental): Six hundred mg of rifampicin (2 tablets of 300mg Rifadine; Sanofi, Belgium) will be administered once daily on days 7 through 13.
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Voriconazole
  Other Names: Vfend
  Arms: Voriconazole
Drug: Rifampin
  Other Names: Rifadin; Rifadine
  Arms: Rifampin

SUMMARY:
Single center, open label crossover study with 2 treatment phases in healthy volunteers.

The potential of phenotypic drug probes to predict drug-drug interactions between tacrolimus, voriconazole and rifampin will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age over 18 years
* Written informed consent

Exclusion Criteria:

* Female
* Medical comorbidities
* Use of concomitant medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in tacrolimus area under the curve | 2 weeks
  assessed twice: once after each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dirk RJ Kuypers, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium